CLINICAL TRIAL: NCT03831464
Title: Metformin as RenoProtector in Non-Diabetic Patients With Progressive Chronic Kidney Disease (CKD Stages 2, 3A and 3B): a Multi-centre, Practice-oriented, Repurposing, Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Metformin as RenoProtector of Progressive Kidney Disease
Acronym: RenoMet
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Prof Dr. Marc De Broe, Prof Dr., Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RenoMet
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Diseases
Keywords: CKD; Metformin; Renoprotector
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: A multi-center, practice-oriented, repurposing, double-blinded, placebo-controlled, randomized clinical trial. The RenoMet trial is repurposing an already approved agent (Metformin , Glucophage SR) in a new indication (renoprotection) in a new class of patients (chronic kidney disease patients CKD 2, 3A, 3B and including patients with renal transplant for more than 3 years),
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin treatment group (Experimental)
  Interventions: Drug: Metformin Hydrochloride
- Placebo control group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin Hydrochloride — The intervention will consist in IMP treatment during 30 months with half of the patients treated with Metformin Glucophage SR. Tablets of 500mg will be used at a dose of 2x500mg preferably taken during the evening meal.
  During the first month of the trial a dose of 1x500mg will be used in order to avoid as much as possible some well-known mainly gastrointestinal side effects of metformin treatment .
  Arms: Metformin treatment group
Drug: Placebo Oral Tablet — The intervention will consist in IMP treatment during 30 months with half of the patients treated with matched placebo. Tablets of 500mg will be used at a dose of 2x500mg preferably taken during the evening meal.
  Arms: Placebo control group

SUMMARY:
A multi-center, practice-oriented, repurposing, double-blinded, placebo-controlled, randomized clinical trial. The RenoMet trial is repurposing an already approved agent (Metformin , Glucophage SR ) in a new indication (renoprotection ) in a new class of patients (chronic kidney disease patients CKD 2, 3A, 3B and including patients with renal transplant for more than 3 years).

DETAILED DESCRIPTION:
The intervention consists in the treatment of patients with progressive kidney disease and blindly randomized to the treatment group with metformin as medication, added to their usual treatment. Metformin is a well-known and cheap medication used for many years and still used as main treatment of type 2 diabetes. In our study, this 'old' product will be used for a 'new' indication, slowing down the progression of CKD. After randomization in the participating renal care clinic, patients in the intervention group will be treated with metformin at a dose of 1000 mg/day (2x500mg) in the evening during 30 months (Metformin - Glucophage SR (Merck KGaA)). During the first month of the trial a dose of 1x500mg will be used in order to avoid as much as possible some well-known mainly gastrointestinal side effects of metformin treatment At each visit during the study period, the metformin medication will be hand over to the patient in a HDPE bottle, closed with a MEMS cap (Medication Event Monitoring System). The MEMS a cap that registers the time and date of each opening (presumed intake of the medication in the bottle).

Patients blindly randomized to the control group will receive placebo treatment (2 tablets per day) also in a MEMS device and will continue to receive usual care. Control patients will have the same data collection.

Follow-up of patients during the entire study period will be the responsibility of the treating nephrologist in the renal care clinic. All patients will have a baseline data collection at study entry (demographics, comorbidities, concomitant medication, clinical parameters, lab results). During the study period of 30 months patients will have follow-up visits at their renal care clinic every four months with collection of follow-up data (concomitant medication, clinical parameters, routine lab results and drug related problems). Extra blood and urine samples will be collected for a centralized second determination of serum creatinine and proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) of both gender
* Seen on a regular base in one of the participating outpatient clinics of renal care with a previous consultation within the last year
* Having a chronic kidney disease (including having a transplant kidney for more than 3 years) with:

  * a CKD stage 2, 3A or 3B (i.e. with estimated glomerular filtration rate (eGFR) between 30 and 70 ml/min/1.73m2) at the time of the baseline visit
  * showing a decline of eGFR between 3.0 and 20.0 ml/min/year determined using at least three determinations of eGFR (CKD-Epi formula) whereby the oldest one should be from more than 1 year ago and the most recent will be the one of the baseline visit. For transplant patients the decline will be based on serum creatinine values determined during the preceding 24 months. For all other patients, the decline will be based on values determined within the last five years

Exclusion Criteria:

1. Illiteracy: patients not knowing how to read or write
2. Patients not able to communicate in Dutch or French
3. Patients with mental deterioration, incapable to give informed consent and to understand the safety instructions of the study (at the discretion of the treating nephrologist)
4. Patients with one of the following clinical problems:

   * Patients with nephrotic syndrome
   * Patients showing a fast decline of renal function (more than 20 ml/min/year) during the preceding five years
   * Diabetes mellitus (any type: 1, 2, Maturity Onset Diabetes of the Young (MODY), New Onset Diabetes After Transplantation (NODAT)) confirmed by a glycemia level >125 mg/dl (7.0 mmol/L) after a fasting time of 8 hours
   * Patients with a renal transplantation for less than 3 years
   * Patients with multi-organ transplantation
   * History of other solid organ transplantations
   * Chronic obstructive pulmonary disease (COPD) stage Gold IV (Oxygene-dependency)
   * Congestive heart failure (NYHA stage IV)
   * Inflammatory bowel disease (IBD)
   * Stoma
   * Hepatic insufficiency or cirrhosis, acute alcohol intoxication or alcoholism (> 20 glasses of alcoholic beverages per week)
   * History of metabolic diseases (e.g. mitochondrial encephalomyopathy (MELAS), lactic acidosis, stroke-like episodes, etc…)
   * Pregnancy and/or lactating women at the time of recruitment and during the study period
   * Patient with prior use of metformin within the past 12 months (e.g. glucose intolerance, polycystic ovary syndrome, etc…) or with other study medication taken within the framework of another clinical trial
5. Patients showing elevated blood lactate level(s) at the time of recruitment (i.e. a confirmed lactate level ≥ 2.5 mmol/L at baseline and a confirmed lactate level ≥ 2.5 mmol/L after 4 weeks (±1 week)).
6. Patients showing a confirmed (after 3 months) serum bicarbonate level < 22 mmol/L (or < 20 mmol/L if delay of more than 1 hour between sampling and determination)
7. Hypersensitivity to metformin or to any of the excipients listed in section 6.1 of the Glucophage SR SmPC (see Attachment A5 Glucophage SR SmPC)
8. One of the following diseases during the previous 6 months: myocardial infarction, shock, acute problems of decompensated heart failure or respiratory failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reaching a 30% decline of eGFR | Period of 30 months
  Values of serum creatinine obtained from local determination will be used for the calculation of eGFR.

SECONDARY OUTCOMES:
Mortality rate during the investigation period | Period of 30 months
  The time to the event of all-cause mortality will be compared between Metformin and placebo.
Evolution of the renal function | Period of 30 months
  Expressed as the slopes of the 8 eGFR determinations during the study period
Percentage of patients developing end-stage renal disease | Period of 30 months
  The time to development a doubling of serum creatinine or end-stage renal failure will be compared between Metformin and placebo.
Percentage of transplant patients with graft loss | Period of 30 months
  The time to the event of graft loss will be compared in the Transplant group between Metformin and placebo using a log-rank test. Kaplan Meier curves will be used to describe the data graphically.
Evolution of proteinuria | Difference between baseline and study end
  This will be examined by a generalized linear mixed models using baseline measurement and study end measurement.
Evolution of hypertension | Difference between baseline and study end
  This will be examined by a generalized linear mixed models using baseline measurement and study end measurement.
Frequency of Major Adverse Cardiovascular Events | Period of 30 months
  This will be examined by a generalized linear mixed models using baseline measurement and study end measurement. This model will allow inclusion of correcting variables.
Hospitalization during the investigation period | Period of 30 months
  Hospitalization during the investigation period will be studied using a Cox regression with multiple events.
Hospitalization during the investigation period | Period of 30 months
  Total number of hospitalization days will be analyzed using a multiple regression model.
(Serious) Adverse drug events | Period of 30 months
  Number of lactic acidosis events, number of deaths related to lactic acidosis, other adverse events. Reported selected AEs and all SAEs will be summarized using descriptive statistics and a comparison between Metformin and placebo group will be performed.
Evolution of Quality of life | Period of 30 months
  During the study period (area under the curve as well as difference between baseline and study end) of the utility Qol score of the EQ-5D-5L questionnaire. Quality of life as measured during the follow-up visits as well as the evolution of Qol during the trial will be compared between Metformin and placebo group.

CONTACTS AND LOCATIONS:
Locations (19):
- Belgium (19):
  - AZ Delta, Roeselare, West-Vlaanderen
  - OLVZ Aalst, Aalst
  - Epicura Ath, Ath
  - Epicura Baudour, Baudour
  - Imelda Ziekenhuis Bonheiden, Bonheiden
  - CHU Brugmann, Brussels
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Antwerp University Hospital, Edegem
  - Ghent University Hospital, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Centre Hospitalier Régional de la Citadelle, Liège
  - Centre Hospitalier Universitaire Liège (CHU Liège), Liège
  - Centre Hospitalier Régional de Namur, Namur
  - AZ Nikolaas, Sint-Niklaas
  - Centre Hospitalier de Wallonie Picarde, Tournai
  - AZ Turnhout, Turnhout
  - CHR Verviers, Verviers

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240